CLINICAL TRIAL: NCT05391451
Title: Clinical Efficacy of the Quadratus Lumborum Block for Analgesia in Kidney Transplant Surgery
Brief Title: New Approach of Loco Regional Analgesia in Kidney Transplant
Acronym: CARRENAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PO21061
Record Dates: First submitted 2022-05-19; First posted 2022-05-26 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Diseases
Keywords: Analgesia; Chronic kidney disease; Renal Transplant
MeSH Terms: conditions — Renal Insufficiency, Chronic; Agnosia | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus lumborum block (QLB) group (Experimental)
  Interventions: Procedure: efficacy of quadratus lumborum block in post-operative analgesia in kidney transplant surgery
- Control group (Active Comparator)
  Interventions: Procedure: general anesthesia

INTERVENTIONS:
Procedure: efficacy of quadratus lumborum block in post-operative analgesia in kidney transplant surgery — no premedication for anxiolytic purposes before surgery. Cimetidin 200mg can be administrated for Mendelson syndrome prevention. After general anesthesia induction, echo-guided quadratus lumborum block is performed by applying 20ml of levobupivacaine
  Arms: Quadratus lumborum block (QLB) group
Procedure: general anesthesia — general anesthesia is the current technique for kidney transplant surgery. The protocol involves the combination of several drugs: Propofol, Remifentanil, Ketamin, Atracurium or Cisatracurium. Curarization monitoring is systematic.
  Arms: Control group

SUMMARY:
Kidney transplant is considered as a moderate painful surgery. Unfortunately, patients with chronic kidney disease are not able to degrade opioid drugs and are therefore most likely to be subjected to the secondary effects of their consumption. Current strategies aim to find pain relief substitutes in order to decrease the use of opioids, specially after surgery, during patient recovery. Loco-regional analgesia consists of administering local anesthesic directly in specific nerves and is being used in several surgical procedures. In various abdominal surgeries, a loco-regional analgesia called "tranversus abdominis Plane Block" has been associated with decreased morphine consumption and better post-operative conditions. In kidney transplant, the definitive efficacy of this loco-regional analgesia is not established, due to controversial clinical results.

The goal of our study is to test the analgesia advantage of a variant of the Tranversus Abdominis Plane Block, called Quadratus lumborum block, which targets a muscle called quadratus lumborum, in association with general anesthesia, on post-surgery recovery and opioid intake.

DETAILED DESCRIPTION:
Post-operative pain after a kidney transplant can be moderate to severe, but analgesic options are limited. Clearance of the active metabolite of morphin is low in patients with chronic kidney disease, which imposes a strict monitoring of morphin administration. Therefore pain control is difficult and non-optimal.

Reducing both pain and opioid consumption during the per and post operative periods constitutes a major stake, and involves the use of locoregional anesthesia techniques.

The recent literature recommends the realization of a transversus abdominal plane block, despite contradictory results concerning the expected effect.

Even though peridural analgesia remains the gold standard in many types of surgeries, it is not recommended in case of renal transplant due to multiple secondary effects.

The quadratus lumborum bloc echoguid is a recent technique of locoregional analgesia, used in lower abdominal surgeries (appendicectomy, césarian, digestive resection, …) "because of a prolonged duration of action and a sensitive anesthesia spreading" (which provides a much wider field of analgesia?). This technique is not described for the kidney transplant surgery.

This type of bloc will be realized after the induction of general anesthesia. The patient will be positioned in dorsal decubitus with a lumbar block or in left lateral decubitus to expose the iliac fossa and the right flan. After echographia landmark, a solution of local anesthesic will be place in contact of the quadratus lumborum muscle, into the median beam, to obtain a crescent moon image, sign of the good spreading of the local anesthesic.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for kidney transplant surgery at the CHU de Reims
* Patients agreeing to participate in the research and having signed the informed consent
* Adult patients
* Patients affiliated to a social security scheme

Exclusion Criteria:

* Legally protected
* Known allergy to local anesthetics used
* Manifest polyneuropathy
* ASA score > 4
* Pregnancy, breastfeeding
* Contraindications to QLB
* Technique refusal
* Previous kidney transplant
* History of major abdominal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-10-23 (Actual)

PRIMARY OUTCOMES:
consumption of morphine | Day 1
  Total consumption of morphine during the first day after surgery

SECONDARY OUTCOMES:
consumption of ULTIVA | Day 0
  Total consumption of ULTIVA during the surgery
Pain evaluation | Hour 1
  Pain evaluation at various timepoints by Visual Analog Scale
Pain evaluation | Hour 2
  Pain evaluation at various timepoints by Visual Analog Scale
Pain evaluation | Hour 6
  Pain evaluation at various timepoints by Visual Analog Scale
Pain evaluation | Hour 12
  Pain evaluation at various timepoints by Visual Analog Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France